CLINICAL TRIAL: NCT02079532
Title: An Open-label Study to Evaluate the Safety of MabThera, and Its Effect on Treatment Response, in Patients With Rheumatoid Arthritis Following Inadequate Response to a Single Anti-TNF Agent
Brief Title: A Study of MabThera (Rituximab) in Patients With Rheumatoid Arthritis Who Have Had an Inadequate Response to a Single Anti-TNF Inhibitor
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML19070
Record Dates: First submitted 2014-03-04; First posted 2014-03-05 (Estimated); Results first posted 2015-06-09 (Estimated); Last update posted 2016-07-29 (Estimated); Status verified 2016-06

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Rituximab

ARMS (1):
- MabThera (Rituximab) (Experimental)
  Interventions: Drug: rituximab [MabThera]

INTERVENTIONS:
Drug: rituximab [MabThera] — 1 g was given by intravenous infusion on Days 1 and 15

SUMMARY:
This study will evaluate the efficacy and safety of MabThera in patients with active rheumatoid arthritis who have had an inadequate response to one prior anti-TNF alpha inhibitor. MabThera-naive patients will be stratified into 3 arms, according to previous inadequate response to a)etanercept, b)infliximab or c)adalimumab. Patients will be treated with MabThera (1g infusion) on day 1 and day 15, and will continue their basic methotrexate therapy. The anticipated time on study treatment is 2+ years, and the target sample size is 100-500 individuals.

ELIGIBILITY:
Inclusion Criteria:

* adult patients, 18-75 years of age;
* rheumatoid arthritis for >=6 months;
* previous inadequate response to a single anti-TNF alpha inhibitor;
* methotrexate at a stable dose range 7.5-25 mg/week.

Exclusion Criteria:

* other chronic inflammatory articular disease or systemic autoimmune disease;
* previous treatment with MabThera or intolerance to MabThera;
* corticosteroids>=10 mg/day prednisolone within last 2 weeks, or corticosteroids at unstable doses within last 2 weeks;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 302 (Actual)
Dates: Start 2006-11; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Chair — Hoffmann-La Roche
Locations (56):
- Germany (56):
  - Bad Abbach
  - Bad Aibling
  - Bad Bramstedt
  - Bamberg
  - Berlin
  - Bonn
  - Bremen
  - Cologne
  - Cuxhaven
  - Damp
  - Donaueschingen
  - Dresden
  - Düsseldorf
  - Erfurt
  - Erlangen
  - Essen
  - Frankfurt am Main
  - Freiburg im Breisgau
  - Fulda
  - Giessen
  - Gommern
  - Göttingen
  - Hagen
  - Halle
  - Hamburg
  - Hanover
  - Heidelberg
  - Herne
  - Hofheim
  - Homburg/saar
  - Jena
  - Karlsruhe
  - Ludwigshafen
  - Mainz
  - Mittelherwigsdorf
  - Mönchengladbach
  - München
  - Münster
  - Naunhof
  - Oldenburg
  - Osnabrück
  - Pirna
  - Ratingen
  - Rostock
  - Schwerte
  - Sendenhorst
  - Stuttgart
  - Treuenbrietzen
  - Trier
  - Tübingen
  - Ulm
  - Wiesbaden
  - Wuppertal
  - Würselen
  - Würzburg
  - Zeven

RESULTS

PARTICIPANT FLOW:
Groups:
- Rituximab Plus Methotrexate (MTX): Participants received rituximab, 1 gram (g), intravenously (IV), and methylprednisolone 100 mg, IV, on Days 1 and 15. Participants should have also been receiving MTX as mandatory background therapy. MTX was to have been started at least 3 months prior to the first infusion and must have been given at stable doses for at least 4 weeks prior to the first infusion.
Period: Overall Study
Arm/Group | Rituximab Plus Methotrexate (MTX)
Started | 302
Completed | 273
Not Completed | 29
Not completed — Adverse Event | 7
Not completed — Additional or changed therapy | 2
Not completed — Lack of Efficacy | 9
Not completed — Protocol Violation | 3
Not completed — Withdrawal by Subject | 1
Not completed — Administrative problems | 1
Not completed — Inclusion into ReFIRST | 3
Not completed — Other | 3

BASELINE CHARACTERISTICS:
Population: Safety population: all participants who received at least 1 dose of trial medication and had at least 1 safety follow-up.
Groups:
- Rituximab + MTX: Participants received rituximab, 1 g, IV, and methylprednisolone 100 mg, IV, on Days 1 and 15. Participants should have also been receiving MTX as mandatory background therapy. MTX was to have been started at least 3 months prior to the first infusion and must have been given at stable doses for at least 4 weeks prior to the first infusion.
Arm/Group | Rituximab + MTX
Number analyzed (Participants) | 302
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.4 (18.77)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 228
  Male | 74
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 301
  Asian | 1

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Week 24 in Disease Activity Score Based on 28-Joint Count (DAS28)
Description: The DAS28 consists of swollen joint count (SJC) and tender joint count (TJC) measurements, the erythrocyte sedimentation rate (ESR) in millimeters per hour (mm/hr), and the Patient's Global Assessment of Disease Activity (participant-ated rheumatoid arthritis [RA] activity assessment) with transformed scores ranging 0 to 10; higher scores indicated greater affectation due to disease activity). DAS28 less than or equal to (≤)3.2 equals (=) low disease activity, DAS28 greater than (>)3.2 to 5.1 = moderate to high disease activity.
Time Frame: Week 24
Population: Intent to Treat (ITT) population: all participants who signed informed consent, received at least 1 dose of study drug, and where DAS28 was measured at least once under study medication (Weeks 8, 16, or 24 or unscheduled or withdrawal visit up to Week 24); those with no RA or no DAS28 score at screening were excluded, regardless if treated or not.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Rituximab + MTX
Number analyzed (Participants) | 291
scores on a scale | -1.56 (1.40)

2. Secondary Outcome: DAS28 Score
Description: The DAS28 consists of SJC and TJC measurements, the ESR in mm/hr, and the Patient's Global Assessment of Disease Activity (participant-rated RA assessment) with transformed scores ranging 0 to 10; higher scores indicated greater affectation due to disease activity). DAS28 ≤3.2 = low disease activity, DAS28 >3.2 to 5.1 = moderate to high disease activity.
Time Frame: Screening and Weeks 8, 16, and 24
Population: ITT population; n (number) = number of participants assessed at a given visit.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Rituximab + MTX
Number analyzed (Participants) | 291
scores on a scale
  Screening (n=291) | 5.87 (1.05)
  Week 8 (n=277) | 4.57 (1.30)
  Week 16 (n=271) | 4.17 (1.31)
  Week 24 (n=266) | 4.30 (1.47)

3. Secondary Outcome: Percentage of Participants With European League Against Rheumatism (EULAR) Response of Good or Moderate
Description: The DAS28-based EULAR response criteria were used to measure individual responses as none, good, and moderate, depending on the extent of change from baseline and the level of disease activity reached. Good responders experienced a change from baseline of >1.2 with a DAS28 score ≤3.2 and moderate responders experienced a change from baseline >1.2 with DAS28 >3.2 to ≤5.1 or a change from baseline >0.6 to ≤1.2 with a DAS28 score of ≤5.1.
Time Frame: Weeks 8, 16, and 24
Population: ITT population; n=number of participants assessed at a given visit
Measure: Number; unit: percentage of participants
Arm/Group | Rituximab + MTX
Number analyzed (Participants) | 291
percentage of participants
  Week 8 (n=172) | 59.1
  Week 16 (n=198) | 68.0
  Week 24 (n=188) | 64.6

4. Secondary Outcome: Percentage of Participants With Low Disease Activity (DAS28 ≤3.2) at Week 24
Description: Percentage of participants with low disease activity defined as DAS28 ≤3.2 at follow-up Week 24. The DAS28 consists of SJC and TJC measurements, the ESR in mm/hr, and the Patient's Global Assessment of Disease Activity (participant rated arthritis activity assessment) with transformed scores ranging 0 to 10; higher scores indicated greater affectation due to disease activity).
Time Frame: Week 24
Population: ITT population
Measure: Number; unit: percentage of participants
Arm/Group | Rituximab + MTX
Number analyzed (Participants) | 291
percentage of participants | 21.6

5. Secondary Outcome: Percentage of Participants Achieving Remission (DAS28 <2.6) at Week 24
Description: Percentage of participants with remission defined as DAS28 <2.6 at follow-up Week 24. The DAS28 consists of SJC and TJC measurements, the ESR in mm/hr, and the Patient's Global Assessment of Disease Activity (participant rated arthritis activity assessment) with transformed scores ranging 0 to 10; higher scores indicated greater affectation due to disease activity). DAS28 ≤3.2 = low disease activity, DAS28 >3.2 to 5.1 = moderate to high disease activity.
Time Frame: Week 24
Population: ITT population
Measure: Number; unit: percentage of participants
Arm/Group | Rituximab + MTX
Number analyzed (Participants) | 291
percentage of participants | 11.7

6. Secondary Outcome: Percentage of Participants Achieving a Response By EULAR Category
Description: Percentage of participants achieving a response by EULAR category, including 'moderate', 'good', or no response at follow-up Weeks 8, 16, and 24. The DAS28-based EULAR response criteria were used to measure individual response as none, good, and moderate, depending on the extent of change from baseline and the level of disease activity reached. Good responders had a change from baseline >1.2 with a DAS28 score ≤ 3.2; moderate responders had a change from baseline >1.2 with a DAS28 score of >3.2 to ≤5.1 or a change from baseline >0.6 to ≤1.2 with a DAS28 score of ≤5.1; non-responders had a change from baseline ≤0.6 or change from baseline >0.6 and ≤1.2 with a DAS28 score of >5.1.
Time Frame: Weeks 8, 16, and 24
Population: ITT population
Measure: Number; unit: percentage of participants
Arm/Group | Rituximab + MTX
Number analyzed (Participants) | 291
percentage of participants
  Moderate response, Week 8 | 45.4
  Moderate response, Week 16 | 44.3
  Moderate response, Week 24 | 44.0
  Good response, Week 8 | 13.7
  Good response, Week 16 | 23.7
  Good response, Week 24 | 20.6
  No response, Week 8 | 36.1
  No response, Week 16 | 25.1
  No response, Week 24 | 26.8

7. Secondary Outcome: Health Assessment Questionnaire - Disability Index (HAQ-DI) Score
Description: The HAQ-DI score consists of questions referring to 8 categories: dressing/grooming, arising, eating, walking, hygiene, reach, grip, and common daily activities. For each of the categories, participants reported the amount of difficulty they had in performing 2 or 3 specific sub-category items. The standard disability score was calculated from the 8 categories by dividing the sum of the individual categories by the number of categories answered, yielding a score from 0 (without any difficulty) to 3 (unable to do).
Time Frame: Screening and Weeks 8, 16, and 24
Population: ITT population; n=number of participants assessed at a given visit.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Rituximab + MTX
Number analyzed (Participants) | 291
scores on a scale
  Screening (n=288) | 1.60 (0.67)
  Week 8 (n=286) | 1.43 (0.66)
  Week 16 (n=276) | 1.33 (0.66)
  Week 24 (n=269) | 1.32 (0.70)

8. Secondary Outcome: Functional Assessment of Chronic Illness Therapy - Fatigue (FACIT-F) Score
Description: The FACIT fatigue scale is base on a 13-item questionnaire to assess the therapy-induced fatigue. Participants were requested to score each question on a scale ranging from 0 (best) to 4 (worst). The scoring system of the FACIT fatigue scale adds up to a total scale ranging from 0 (best) to 52 (worst). The assessment was originally developed for chronic illnesses and is now validated for patients with rheumatoid arthritis (RA). The questionnaire was provided in a German translation.
Time Frame: Screening and Weeks 8, 16, and 24
Population: ITT population; n=number of participants assessed at a given visit.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Rituximab + MTX
Number analyzed (Participants) | 291
scores on a scale
  Screening (n=286) | 23.81 (11.35)
  Week 8 (n=282) | 20.87 (11.14)
  Week 16 (n=272) | 18.92 (11.46)
  Week 24 (n=262) | 18.53 (11.48)

9. Secondary Outcome: Short-Form 36 (SF-36) Physical Composite Scores (PCS) and Mental Composite Scores (MCS)
Description: The SF-36 is a multi-purpose, short-form health survey with 36 questions. It yields an 8-scale profile of functional health and well-being scores (domains) as well as psychometrically based physical and mental health summary measures. The SF-36 taps 8 health concepts: physical functioning, bodily pain, physical role functioning, emotional role functioning, emotional well-being, social functioning, vitality, and general health perceptions. The 8 scales are further summarized to 2 distinct higher-ordered clusters: the physical and mental composite t-scores (PCS and MCS). The range for all 8 domains as well as for the composite t-scores is from 0 to 100 with 100 as best possible health status and 0 as worst health status.
Time Frame: Screening and Weeks 8, 16, and 24
Population: ITT population; n=number of participants assessed at a given visit.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Rituximab + MTX
Number analyzed (Participants) | 291
scores on a scale
  PCS, Screening (n=287) | 30.97 (8.14)
  PCS, Week 8 (n=279) | 34.24 (8.56)
  PCS, Week 16 (n=270) | 35.92 (8.43)
  PCS, Week 24 (n=264) | 36.36 (9.00)
  MCS, Screening (n=287) | 40.88 (13.16)
  MCS, Week 8 (n=279) | 43.50 (12.31)
  MCS, Week 16 (n=270) | 45.17 (12.32)
  MCS, Week 24 (n=264) | 44.92 (13.13)

10. Secondary Outcome: SF-36 Domain Scores
Description: The SF-36 is a multi-purpose, short-form health survey with 36 questions. It yields an 8-scale profile of functional health and well-being scores (domains) as well as psychometrically based physical and mental health summary measures. The SF-36 taps 8 health concepts: physical functioning, bodily pain, physical role functioning, emotional role functioning, emotional well-being, social functioning, vitality, and general health perceptions. The 8 scales are further summarized to two distinct higher-ordered clusters: the physical and mental composite t-scores (PCS and MCS). The range for all 8 domains as well as for the composite t-scores is from 0 to 100 with 100 as best possible health status and 0 as worst health status.
Time Frame: Screening and Weeks 8, 16, and 24
Population: ITT population; n=number of participants assessed at a given visit.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Rituximab + MTX
Number analyzed (Participants) | 291
scores on a scale
  Physical functioning, Screening (n=289) | 39.04 (24.83)
  Physical functioning, Week 8 (n=284) | 43.60 (24.50)
  Physical functioning, Week 16 (n=276) | 44.64 (25.13)
  Physical functioning, Week 24 (n=268) | 47.37 (26.19)
  Bodily pain, Screening (n=290) | 25.94 (17.75)
  Bodily pain, Week 8 (n=285) | 37.24 (19.00)
  Bodily pain, Week 16 (n=275) | 44.25 (21.60)
  Bodily pain, Week 24 (n=267) | 44.06 (22.13)
  Physical role functioning, Screening (n=290) | 35.11 (22.42)
  Physical role functioning, Week 8 (n=284) | 43.72 (23.95)
  Physical role functioning, Week 16 (n=276) | 48.37 (23.48)
  Physical role functioning, Week 24 (n=269) | 49.63 (25.04)
  Emotional role functioning, Screening (n=289) | 52.77 (31.23)
  Emotional role functioning, Week 8 (n=282) | 59.13 (27.26)
  Emotional role functioning, Week 16 (n=276) | 62.41 (27.57)
  Emotional role functioning, Week 24 (n=268) | 61.29 (27.98)
  Emotional well-being, Screening (n=289) | 56.11 (20.07)
  Emotional well-being, Week 8 (n=285) | 60.43 (19.82)
  Emotional well-being, Week 16 (n=276) | 63.02 (20.51)
  Emotional well-being, Week 24 (n=268) | 64.03 (21.03)
  Social functioning, Screening (n=291) | 56.62 (27.23)
  Social functioning, Week 8 (n=285) | 64.04 (25.87)
  Social functioning, Week 16 (n=277) | 65.93 (26.10)
  Social functioning, Week 24 (n=270) | 66.99 (28.11)
  Vitality, Screening (n=290) | 38.49 (19.41)
  Vitality, Week 8 (n=285) | 43.42 (19.76)
  Vitality, Week 16 (n=276) | 48.25 (20.32)
  Vitality, Week 24 (n=268) | 48.22 (20.75)
  General health perceptions, Screening (n=291) | 39.14 (14.49)
  General health perceptions, Week 8 (n=285) | 45.61 (15.06)
  General health perceptions, Week 16 (n=272) | 48.54 (17.16)
  General health perceptions, Week 24 (n=269) | 48.30 (17.53)

11. Secondary Outcome: Percentage of Participants Achieving American College of Rheumatology (ACR) 20 Percent (%), 50% or 70% Response (ACR20/ACR50/ACR70)
Description: ACR20/50/70 response: ≥20%, ≥50%, or ≥70% improvement, respectively, in tender or swollen joint counts and ≥20%, ≥50%, or ≥70% improvement, respectively, in 3 of the following 5 criteria: 1) Physician's Global Assessment of Disease Activity, 2) Patient's Global Assessment of Disease Activity, 3) Patient's Assessment of Pain, 4) participant assessment of functional disability via a HAQ-DI, and 5) C-reactive protein or ESR at each visit.
Time Frame: Weeks 8, 16, and 24
Population: ITT population
Measure: Number; unit: percentage of participants
Arm/Group | Rituximab + MTX
Number analyzed (Participants) | 291
percentage of participants
  ACR20, Week 8 | 38.8
  ACR20, Week 16 | 47.8
  ACR20, Week 24 | 46.4
  ACR50, Week 8 | 13.7
  ACR50, Week 16 | 19.9
  ACR50, Week 24 | 24.4
  ACR70, Week 8 | 2.7
  ACR70, Week 16 | 8.2
  ACR70, Week 24 | 10.0

12. Secondary Outcome: Swollen Joint Count (SJC)
Description: The 28 joints to be assessed for tenderness and swelling were shoulder, elbow, wrist, metacarpophalangeal (MCP) joints 1-5, proximal interphalangeal (PIP) joints 1-5, and knee on both sides of the body. The sum of swollen joints, each, ranged from 0 to 28 with 0 as best possible health status and 28 as worst health status.
Time Frame: Screening and Weeks 8, 16, and 24
Population: ITT population; n=number of participants assessed at a given visit.
Measure: Mean (Standard Deviation); unit: swollen joints
Arm/Group | Rituximab + MTX
Number analyzed (Participants) | 291
swollen joints
  Screening (n=291) | 10.01 (5.34)
  Week 8 (n=288) | 5.16 (4.73)
  Week 16 (n=282) | 4.22 (4.07)
  Week 24 (n=272) | 4.70 (4.67)

13. Secondary Outcome: Tender Joint Count (TJC)
Description: The 28 joints to be assessed for tenderness and swelling were shoulder, elbow, wrist, metacarpophalangeal (MCP) joints 1-5, proximal interphalangeal (PIP) joints 1-5, and knee on both sides of the body. The sum of tender joints ranged from 0 to 28 with 0 as best possible health status and 28 as worst health status.
Time Frame: Screening and Weeks 8, 16, and 24
Population: ITT population; n=number of participants assessed at a given visit.
Measure: Mean (Standard Deviation); unit: tender joints
Arm/Group | Rituximab + MTX
Number analyzed (Participants) | 291
tender joints
  Screening (n=291) | 12.62 (6.31)
  Week 8 (n=288) | 7.53 (6.71)
  Week 16 (n=282) | 6.04 (6.31)
  Week 24 (n=272) | 6.41 (6.37)

14. Secondary Outcome: Physician's Global Assessment of Disease Activity
Description: Physicians assessed the disease (RA) activity on a 100 mm horizontal VAS. The left-hand extreme of the line (0 mm) was described as "no disease activity" (symptom-free and no arthritis symptoms) and the right hand extreme (100 mm) as "maximum disease activity" (maximum arthritis disease activity).
Time Frame: Screening and Weeks 8, 16, and 24
Population: ITT population; n=number of participants assessed at a given visit.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Rituximab + MTX
Number analyzed (Participants) | 291
mm
  Screening (n=291) | 63.99 (15.40)
  Week 8 (n=286) | 39.20 (19.85)
  Week 16 (n=280) | 33.03 (19.96)
  Week 24 (n=271) | 35.75 (23.92)

15. Secondary Outcome: Patient's Assessment of Disease Activity
Description: Participants were to assess the disease (RA) activity on a 100 mm horizontal VAS. The left-hand extreme of the line (0 mm) was described as "no disease activity" (symptom-free and no arthritis symptoms) and the right hand extreme (100 mm) as "maximum disease activity" (maximum arthritis disease activity).
Time Frame: Screening and Weeks 8, 16, and 24
Population: ITT population; n=number of participants assessed at a given visit.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Rituximab + MTX
Number analyzed (Participants) | 291
mm
  Screening (n=291) | 63.49 (20.88)
  Week 8 (n=286) | 46.19 (23.51)
  Week 16 (n=278) | 41.25 (24.99)
  Week 24 (n=270) | 41.47 (25.50)

16. Secondary Outcome: Patient's Assessment of Pain
Description: Participants were to assess their current level of pain on a 100 mm horizontal VAS. The left-hand extreme of the line (0 mm) was described as "no pain" and the right-hand (100 mm) as "unbearable pain".
Time Frame: Screening and Weeks 8, 16, and 24
Population: ITT population; n=number of participants assessed at a given visit.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Rituximab + MTX
Number analyzed (Participants) | 291
mm
  Screening (n=291) | 62.78 (20.80)
  Week 8 (n=287) | 47.30 (23.26)
  Week 16 (n=276) | 42.11 (25.14)
  Week 24 (n=269) | 41.76 (25.52)

17. Secondary Outcome: C-Reactive Protein (CRP)
Description: Mean CRP as measured as an acute phase reactant by mg per deciliter (mg/dL) at screening, Days 1 and 15, and Weeks 8, 16, and 24.
Time Frame: Screening, Days 1 and 15, and Weeks 8, 16, and 24
Population: ITT population; n=number of participants assessed at a given visit.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Rituximab + MTX
Number analyzed (Participants) | 289
mg/dL
  Screening (n=289) | 1.82 (2.35)
  Day 1 (n=233) | 1.60 (1.96)
  Day 15 (n=286) | 1.81 (2.27)
  Week 8 (n=283) | 1.31 (1.44)
  Week 16 (n=281) | 1.21 (1.65)
  Week 24 (n=269) | 1.30 (1.77)

18. Secondary Outcome: Erythrocyte Sedimentation Rate (ESR)
Description: Mean ESR, as an acute phase reactant, measured in mm/hr at screening, Days 1 and 15, and Weeks 8, 16, and 24.
Time Frame: Screening, Days 1 and 15, and Weeks 8, 16, and 24
Population: ITT population; n=number of participants assessed at a given visit.
Measure: Mean (Standard Deviation); unit: mm/hr
Arm/Group | Rituximab + MTX
Number analyzed (Participants) | 291
mm/hr
  Screening (n=291) | 30.20 (20.56)
  Day 1 (n=225) | 28.07 (19.51)
  Day 15 (n=277) | 30.61 (21.46)
  Week 8 (n=279) | 24.85 (16.68)
  Week 16 (n=276) | 22.28 (16.58)
  Week 24 (n=268) | 23.64 (17.36)

19. Secondary Outcome: Rheumatoid Factor (RF)
Description: Mean RF as measured by international unit per milliliter (IU/mL) at screening and Weeks 8, 16, and 24.
Time Frame: Screening and Weeks 8, 16, and 24
Population: ITT population; n=number of participants assessed at a given visit.
Measure: Mean (Standard Deviation); unit: IU/mL
Arm/Group | Rituximab + MTX
Number analyzed (Participants) | 279
IU/mL
  Screening (n=279) | 178.23 (352.61)
  Week 8 (n=255) | 109.84 (213.32)
  Week 16 (n=259) | 88.22 (174.99)
  Week 24 (n=258) | 87.52 (187.94)

ADVERSE EVENTS:
Time Frame: From first dose of study drug up to 24 weeks of follow up.
Description: Note that available data included a summary of events by system organ class only, no data provided by preferred term.
Arm/Group | Rituximab + MTX
Serious Adverse Events (participants affected / at risk) | 36/302
Other Adverse Events (participants affected / at risk) | 62/302
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Rituximab + MTX (N=302)
Musculoskeletal and connective tissue disorders (Musculoskeletal and connective tissue disorders) | 9
Infections and infestations (Infections and infestations) | 7
Injury, poisoning and procedural complications (Injury, poisoning and procedural complications) | 7
Gastrointestinal disorders (Gastrointestinal disorders) | 5
Cardiac disorders (Cardiac disorders) | 3
General disorders and administration site conditions (General disorders) | 2
Neoplasms benign, malignant and unspecified (incl cysts and polyps) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Nervous system disorders (Nervous system disorders) | 2
Ear and labyrinth disorders (Ear and labyrinth disorders) | 1
Endocrine disorders (Endocrine disorders) | 1
Immune system disorders (Immune system disorders) | 1
Investigations (Investigations) | 1
Metabolism and nutrition disorders (Metabolism and nutrition disorders) | 1
Psychiatric disorders (Psychiatric disorders) | 1
Renal and urinary disorders (Renal and urinary disorders) | 1
Reproductive system and breast disorders (Reproductive system and breast disorders) | 1
Skin and subcutaneous tissue disorders (Skin and subcutaneous tissue disorders) | 1
Vascular disorders (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Rituximab + MTX (N=302)
Nasopharyngitis (Infections and infestations) | 37
Cough (Respiratory, thoracic and mediastinal disorders) | 19
Hypertension (Vascular disorders) | 17

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.